CLINICAL TRIAL: NCT01745848
Title: Effect of Roflumilast on Systemic Markers of Bone Metabolism and Endothelial Function in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Roflumilast on Markers of Bone Metabolism and Endothelial Function in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jessica Bon Field, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO12060615
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Results first posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Roflumilast; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Drug (Experimental): Roflumilast 500 μcg, once daily, for 30 days
  Interventions: Drug: Roflumilast

INTERVENTIONS:
Drug: Roflumilast
  Other Names: Daxas; Daliresp

SUMMARY:
Our primary hypothesis is that Roflumilast (500 μcg, once daily) will significantly decrease surrogate markers of bone metabolism and early cardiovascular disease in individuals with moderate to severe airflow obstruction and a chronic bronchitis phenotype.

DETAILED DESCRIPTION:
Study participants will be given Roflumilast 500 micrograms daily for 30 days. At baseline, prior to drug administration, blood samples will be collected for analysis of markers of bone metabolism (C-terminal telopeptide of Type I Collagen (CTx), Amino-terminal Propeptide of Type-1 Procollagen (P1NP) and participants will undergo measurement of endothelial function with measurement of brachial flow mediated dilation. After completion of one month of Roflumilast therapy, participants will have a repeat blood collection for measurement of CTx and P1NP and repeat measurement of brachial flow mediated dilation testing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 50 and 70 with a minimum of ten-pack years of tobacco exposure, airflow obstruction (FEV1/FVC < 0.70) with an FEV1 < 70%
* baseline sputum production at least some of the time as reported on the Saint George's Respiratory Questionnaire, and at least one exacerbation within the past year

Exclusion Criteria:

* Subjects with chronic prednisone use, antiresorptive therapy use (bisphosphonates, calcitonin, parathyroid hormone)
* Subjects with a body mass index less than 18 or greater than 34

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Bon Field, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- Emphysema COPD Research Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants enrolled were assigned to the roflumilast group (no control arm of this study).
Groups:
- Roflumilast: Roflumilast 500 μcg, once daily, for 30 days
  Roflumilast
Period: Overall Study
Arm/Group | Roflumilast
Started | 26
Completed | 20
Not Completed | 6
Not completed — Adverse Event | 6

BASELINE CHARACTERISTICS:
Groups:
- Roflumilast: Roflumilast 500 μcg, once daily, for 30 days
Arm/Group | Roflumilast
Number analyzed (Participants) | 26
Age, Continuous [Mean (Full Range); unit: years] | 65.3 [55 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Systemic Markers of Bone Metabolism (C-terminal Peptide of Type 1 Collagen (CTx) and Amino-terminal Propeptide of Type-1 Procollagen (P1NP))
Description: Serum samples were obtained at baseline and after participants took a once daily, 500 mcg roflumilast dose for 30 days. Samples were obtained in the semi-fasting state, processed, and stored for batch analysis at the end of the study. C-terminal peptide of type 1 collagen (CTx), a marker of bone resorption, was analyzed using a commercially available immunoassay (Roche Elecsys 2010 analyzer, Roche Diagnostics, Manheim, Germany). Serum amino-terminal propeptide of type-1 procollagen (P1NP) was measured by ELISA (MyBioSource, San Diego, CA). All assays were performed according to the manufacturers' instructions.
Time Frame: 30 days - measurements at baseline and 30 days
Population: Data were analyzed for the 20 participants completing baseline and follow-up visits after one month on study drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Roflumilast
Number analyzed (Participants) | 20
ng/mL
  change in CTx levels from baseline to 30-days | 0.079 (0.096)
  change in P1NP levels from baseline to 30 days | -101.77 (246.53)

2. Secondary Outcome: Absolute Change From Baseline of Measurements of Brachial Artery Flow Mediated Dilation
Description: Participants had flow mediated dilation of the brachial artery measured at the baseline visit and at the follow-up visit after receiving 30 days of roflumilast 500 mcg daily. An ultrasound probe was placed over the brachial artery and the brachial artery diameter was measured in real time. A blood pressure cuff positioned below the elbow was then inflated to 50 mmHg above systolic pressure for five minutes. After five minutes of occlusion, the blood pressure cuff was released and the brachial artery diameter was again measured in real time. The amount of dilation expressed as the absolute change, in millimeters, from baseline diameter was quantified using the ultrasound images obtained 60 seconds after cuff release.
Time Frame: 30 days - measured at baseline and 30 days
Population: Data were analyzed for the 20 participants completing baseline and follow-up visits after one month on study drug.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Roflumilast
Number analyzed (Participants) | 20
millimeters | 0.335 (4.63)

ADVERSE EVENTS:
Time Frame: 30 days for each participant
Arm/Group | Roflumilast
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 6/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast (N=26)
Gastrointestinal upset (Gastrointestinal disorders) | 3 (3) — diarrhea after starting study drug
Gastrointestinal upset (Gastrointestinal disorders) | 3 (3) — nausea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No